CLINICAL TRIAL: NCT05968495
Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apyx Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APX-23-02
Record Dates: First submitted 2023-07-05; First posted 2023-08-01 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Skin Laxity
Keywords: Renuvion; Helium Plasma
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Renuvion APR System Treatment (Experimental): Subjects are receiving treatment with the Renuvion APR system following power-assisted liposuction in the abdomen per investigator standard of care. Subjects may also have other body areas treated at the same time.
  Interventions: Device: Renuvion APR Handpiece

INTERVENTIONS:
Device: Renuvion APR Handpiece — The Renuvion® APR (Apyx Plasma/RF) handpiece is a sterile, single use electrosurgical (monopolar) device intended to be used in conjunction with a compatible generator for the delivery of radiofrequency energy and helium plasma for cutting, coagulation and ablation of soft tissue during open surgical procedures. Radiofrequency energy is delivered to the handpiece by the generator and used to energize the electrode. When helium gas is passed over the energized electrode, a helium plasma is generated for cutting, coagulation or ablation of soft tissue during open surgical procedures. The compatible generators operate at an adjustable power of up to 40 W (expressed as 0 - 100% where 100% is 40 W) and provide an adjustable helium gas flow of 1 - 5 L/Min. APR Handpiece has a non-extendable electrode to generate helium plasma.

SUMMARY:
This is a prospective, single-center, non-randomized study of up to 5 subjects who are receiving treatment with the Renuvion APR system following power-assisted liposuction in the abdomen per investigator standard of care. Ultrasound images of soft tissue contraction will be taken on abdomen prior to and during the procedure. Measurements of contraction will be calculated from the ultrasound images by an ultrasonographer. All adverse events and expected treatment effects will be documented.

Follow-up photographs and ultrasound images will be captured at D30, D45, D60, D90, D180, D270, & D365.

DETAILED DESCRIPTION:
This is a prospective, single-center, non-randomized study of up to 5 subjects who are receiving treatment with the Renuvion APR system following power-assisted liposuction in the abdomen per investigator standard of care. Subjects may also have other body areas treated at the same time. Demographic information, medical history, and procedure details will be documented. Pre- and post-procedure care are per investigator standard of care and documented. Video may be taken during the procedure.

Ultrasound images of soft tissue contraction will be taken on abdomen prior to and during the procedure. Measurements of contraction will be calculated from the ultrasound images by an ultrasonographer. At baseline, photographs will be taken of the treatment areas. Surface area measurements will be taken of each treatment area prior to study treatment.

Post-procedure care will be as per investigator standard of care and documented. All adverse events and expected treatment effects will be documented.

Follow-up photographs and ultrasound images will be captured at D30, D45, D60, D90, D180, D270, & D365.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for a procedure involving the use of Renuvion for the contraction of subcutaneous soft tissue. Patients undergoing procedures involving Renuvion alone and/or Renuvion following liposuction will be included.
* Patients who have acceptable cardiopulmonary health for outpatient surgery.
* Willing and able to comply with protocol requirements, including obtaining study-required images/photos and assessments, and returning for follow-up visits.
* Willing to release rights for the use of study photos, including in potential publication.
* Able to communicate with the site via video and/or photographs, in the event of a virtual follow-up visit.
* Able to read, understand, sign and date the informed consent document (English only).

Exclusion Criteria:

* BMI of greater than 35.
* Diabetes mellitus with A1C score >7.
* Active cigarette smokers or nicotine vape users.
* History of connective tissue disease (Ehlers Danlos, Cutis Laxa, Pseudoxanthoma Elasticum, Marfan's, etc.)
* Patients who, in the opinion of the investigator, is not an appropriate candidate for the study.
* Patients requiring a concomitant procedure in the Renuvion treatment area that could impact the ultrasound measurements or the effectiveness results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Nichols, Principal Investigator — Investigator; Dan Albershardt, Principal Investigator — Investigator
Locations (1):
- Pearl Plastic Surgery, Olympia, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Renuvion APR System Treatment
Started | 5 (The first study subject was treated on June 12, 2023.)
Completed | 5 (The last subject was treated on September 13, 2023.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: Years] | 48 (44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
BMI [Mean (Full Range); unit: kg/m2] | 30.8 [24.55 to 36.61]

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Contraction From Baseline to Day 365
Description: Percentage of soft tissue contraction measured by an ultrasonographer on baseline ultrasound images compared to follow-up images to quantify the total amount of connective tissue contraction produced by the Renuvion treatment between the skin and the Scarpa's fascia. A negative value indicates greater tissue contraction, while a positive value indicates less tissue contraction.
Time Frame: Baseline, Day 365
Population: During this initial study treatment, the investigators realized the importance of fully expressing the helium from the tissue prior to taking the intra-operative measurements as residual helium expands the subcutaneous tissue, resulting in inaccurate contraction measurements. Due to this discovery and the subsequent change in treatment technique for the remaining subjects, the data for subject 001-BBJ is excluded from the intra-operative data tables and analysis.
Measure: Mean (Standard Deviation); unit: percentage of contraction
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 4
percentage of contraction | -44.0 (17.2)

2. Secondary Outcome: IPR Review
Description: Three experienced, blinded photographic reviewers performed a qualitative analysis/review of pre-treatment and post-treatment sets of images at 90-days, 180-days, 270-days, and 365-days post-treatment compared to baseline for each subject. Images were provided in a blinded and randomized order. Each blinded reviewer choose which set of images were the post-treated Renuvion images of the abdomen. Success was the correct identification of treated abdomen images by at least 2 of the 3 reviewers.
Time Frame: Day 365
Measure: Number; unit: Correctly identified sets of images
Units Other Than Participants: Sets of images analyzed
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 5
Number analyzed (Sets of images analyzed) | 19
Correctly identified sets of images | 18

3. Secondary Outcome: Physician Global Aesthetic Improvement
Description: The Principal Investigator, sub-investigator or qualified clinician delegated by the principal investigator, will complete a PGAIS assessing overall aesthetic improvement in the treatment area.
Time Frame: Day 60, Day 90, Day 180, Day 270, Day 365
Population: One subject missed the D90 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 5
Participants
  Day 60: Worse | 0
  Day 60: No change | 0
  Day 60: Improved, Much Improved, Very Much Improved | 5
  Day 90: number analyzed (Participants) | 4
  Day 90: Worse | 0
  Day 90: No change | 0
  Day 90: Improved, Much Improved, Very Much Improved | 4
  Day 180: Worse | 0
  Day 180: No change | 0
  Day 180: Improved, Much Improved, Very Much Improved | 5
  Day 270: Worse | 0
  Day 270: No change | 0
  Day 270: Improved, Much Improved, Very Much Improved | 5
  Day 365: Worse | 0
  Day 365: No change | 0
  Day 365: Improved, Much Improved, Very Much Improved | 5

4. Secondary Outcome: Subject Global Aesthetic Improvement
Description: The subject will complete a SGAIS assessing overall aesthetic improvement in the treatment area.
Time Frame: Day 60, Day 90, Day 180, Day 270, Day 365
Population: One subject missed the D90 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 5
Participants
  Day 60: Worse | 0
  Day 60: No Change | 0
  Day 60: Improved, Much Improved, Very Much Improved | 5
  Day 90: number analyzed (Participants) | 4
  Day 90: Worse | 0
  Day 90: No Change | 0
  Day 90: Improved, Much Improved, Very Much Improved | 4
  Day 180: Worse | 0
  Day 180: No Change | 0
  Day 180: Improved, Much Improved, Very Much Improved | 5
  Day 270: Worse | 0
  Day 270: No Change | 0
  Day 270: Improved, Much Improved, Very Much Improved | 5
  Day 365: Worse | 0
  Day 365: No Change | 0
  Day 365: Improved, Much Improved, Very Much Improved | 5

5. Secondary Outcome: Patient Satisfaction
Description: The subject will complete a Patient Satisfaction Questionnaire (PSQ)
Time Frame: Day 180, Day 270, Day 365
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 5
Participants
  Characterize Satisfaction with Procedure: Satisfied (Very, Satisfied, or Slightly) | 5
  Noticed improvement in how abdomen looks | 5
  Recommends Procedure to Friends and Family Members | 5
  Improvement Noticed: Improvement in wrinkles | 2
  Improvement Noticed: Less sagging skin | 5
  Improvement Noticed: Smoother skin texture | 3

6. Secondary Outcome: Energy Delivered
Description: Analysis of Energy per surface area was completed for all 5 subjects representing how much energy was delivered to each square centimeter of the abdomen's surface. The general pattern is that the energy per surface area decreases as the surface area of the abdomen increases. Analysis of energy delivered (kJ/cm2)
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: kJ/cm2
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 5
kJ/cm2 | 0.037 (0.012)

ADVERSE EVENTS:
Time Frame: 365 Days
Description: An expected treatment effect was defined as any typical treatment side-effect of Renuvion APR System of mild to moderate severity and lasting up to a typical maximum duration. An adverse event was defined as any new medical problem, or exacerbation of an existing problem, experienced by a subject while enrolled in the study, whether or not it is considered device-related by the investigator.
Arm/Group | Renuvion APR System Treatment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renuvion APR System Treatment (N=5)
Seroma (Surgical and medical procedures) | 3 (3) — These minor seromas were only visible by ultrasound and would have typically gone un-reported had it not been for the ultrasound component of this study.
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 3 (3)
Hypoesthesia/numbness (ETE) (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data produced by this sponsored study is the sole property of Sponsor. Sponsor must be provided with the opportunity to review all Investigator-prepared abstracts, publications, or presentations for a period of thirty (30) days for presentational materials and abstracts and forty-five (45) days for manuscripts.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT05968495/Prot_SAP_000.pdf